CLINICAL TRIAL: NCT01068704
Title: An Open-Label Randomized, Parallel, Two-Arm Phase II Study Comparing BMS-690514 + Letrozole With Lapatinib + Letrozole in Recurrent and Metastatic Breast Cancer Patients Who Are Hormone Receptor Positive Despite HER2 Status And Who Relapsed While Receiving or After Completing Adjuvant Antiendocrine Therapy
Brief Title: Efficacy and Safety of BMS-690514 in Combination With Letrozole to Treat Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA187-016; 2009-016622-13 (EudraCT Number)
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — BMS-690514; Lapatinib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BMS-690514 + Letrozole (Active Comparator)
  Interventions: Drug: BMS-690514; Drug: Letrozole
- Lapatinib + Letrozole (Active Comparator)
  Interventions: Drug: Lapatinib; Drug: Letrozole

INTERVENTIONS:
Drug: BMS-690514 — Tablets, Oral, 200 mg, once daily, ~ 12 months depending on response
  Arms: BMS-690514 + Letrozole
Drug: Lapatinib — Tablets, Oral, 1500 mg, once daily, ~ 12 months depending on response
  Arms: Lapatinib + Letrozole
Drug: Letrozole — Tablets, Oral, 2.5 mg, once daily, ~ 12 months depending on response

SUMMARY:
The purpose of this study is to determine if BMS-690514 + letrozole will be more effective than lapatinib + letrozole in patients who have metastatic hormone receptor positive breast cancer after developing progressive disease immediately following adjuvant antiendocrine therapy

ELIGIBILITY:
Inclusion Criteria:

* Documented invasive breast cancer
* Greater than 10% tumor cells positive for estrogen receptor and/or progesterone receptor
* HER2+ and HER2- (Human Epidermal growth factor Receptor) disease
* Rapid disease progression despite treatment with tamoxifen, anastrozole or exemestane
* ECOG Performance status = 0 or 1

Exclusion Criteria:

* Prior hormonal therapy for metastatic disease
* Prior hormonal therapy with letrozole for adjuvant disease
* Symptomatic brain metastases
* Prior treatment with any tyrosine kinase inhibitor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Rate defined as percentage of subjects with a complete response, partial response, or stable disease for at least 6 months | Every 8 weeks according to CT scan

SECONDARY OUTCOMES:
Progression Free Survival: defined as time to disease progression | Every 8 weeks
Objective Response Rate: defined as percentage of subjects with 'complete response' or 'partial response' | Every 8 weeks
Frequency and severity of adverse events in all subjects | Every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- United States (4):
  - Texas Oncology-Abilene, Abilene, Texas
  - Texas Oncology-Beaumont, Beaumont, Texas
  - Us Oncology Central Pharmacy, Fort Worth, Texas
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
- Argentina (2):
  - Local Institution, La Rioja, La Rioja Province
  - Local Institution, Rosario, Santa Fe Province
- Local Institution, Colima, Colima, Mexico
- Local Institution, Lima, Lima Province, Peru

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx